CLINICAL TRIAL: NCT01684501
Title: Comparing Active and Passive Ankle-foot Prostheses
Status: Completed | Type: Observational
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Other Study IDs: 2010-P-000951
Record Dates: First submitted 2012-09-07; First posted 2012-09-13 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Trans-tibial Amputation
Keywords: prosthesis; amputees; gait

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amputees: Adults with history of traumatic unilateral transtibial amputation

SUMMARY:
The purpose of this study is to perform a biomechanical study of a prototype prosthetic foot and evaluate if it provides a physiological generation of power at the ankle in transtibial amputees. The prosthetic foot is a prototype system that generates power via actuators (i.e. robotic system).

DETAILED DESCRIPTION:
Subjects will be studied during level-ground walking. A camera-based motion capture system will be used to study the biomechanics of motion and evaluate if the pattern of ankle power generation by the prosthetic foot is physiological. In addition, the metabolic cost of ambulation will be monitored during walking at constant speed over a period of several minutes. The data will allow us to assess if the prosthetic foot leads to a decreased metabolic cost of ambulation compared to passive prosthetic feet.

ELIGIBILITY:
Inclusion Criteria:

* weigh more than 200 lbs
* are high level ambulators corresponding to levels E to F of the Special Interest Group of Amputee Medicine (SIGAM) mobility grade
* have the ability to follow multi-step commands.

Exclusion Criteria:

* score level D on the SIGAM mobility grade
* have experienced 1 or more falls in the last month before the study
* have a residual limb length which does not allow for seven inches clearance of bracket attachment for the PowerFoot
* the residual limb must be stable in volume (no change in socket or socket padding in last 6 months) and without pain that limits function
* the sound-side (contralateral) lower extremity must be free of impediments that affect gait, range of motion, or limb muscle activity
* Any diagnosed cardiovascular, pulmonary, neurological, and/ or orthopedic conditions that would interfere with subject participation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with history of traumatic unilateral transtibial amputation
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Ankle power generation | During the session trial (approx 10 minutes)
  Ankle power derived using a camera-based motion capture system during walking

SECONDARY OUTCOMES:
Metabolic cost of ambulation | During the session trial (approx 10 minutes)
  Oxygen consumption during level-ground walking

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No